CLINICAL TRIAL: NCT01319266
Title: An Open-Label, Single-Dose Study to Assess the Pharmacokinetics of the Hydrocodone Bitartrate Extended-Release Tablet (45 mg) in Subjects With Normal Renal Function and Subjects With Varying Degrees of Renal Impairment
Brief Title: A Study to Assess the Pharmacokinetics of the Hydrocodone Extended-Release Tablet (CEP-33237) in Subjects With Normal Renal Function and Subjects With Varying Degrees of Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cephalon (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C33237/1088
Record Dates: First submitted 2011-03-17; First posted 2011-03-21 (Estimated); Last update posted 2012-04-24 (Estimated); Status verified 2012-04

CONDITIONS: Renal Impairment
Keywords: hydrocodone; extended release; pharmacokinetics; renal impairment
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Normal Renal Function (Experimental): Subjects with normal renal function
  Interventions: Drug: Hydrocodone Bitartrate extended-release tablet
- Mild Renal Impairment (Experimental): Subjects with mild renal impairment (defined by an estimated creatinine clearance of > 50 and up to 80 mL/min)
  Interventions: Drug: Hydrocodone Bitartrate extended-release tablet
- Moderate Renal Impairment (Experimental): Subjects with moderate renal impairment (defined by an estimated creatinine clearance of 30-50 mL/min)
  Interventions: Drug: Hydrocodone Bitartrate extended-release tablet
- Severe Renal Impairment (Experimental): Subjects with severe renal impairment (defined by an estimated creatinine clearance of less than 30 mL/min)
  Interventions: Drug: Hydrocodone Bitartrate extended-release tablet
- End Stage Renal Disease (ESRD) (Experimental): Subjects with ESRD (defined as being on hemodialysis for at least 6 months prior to enrollment and be receiving standard in-center dialysis treatments three times a week)
  Interventions: Drug: Hydrocodone Bitartrate extended-release tablet

INTERVENTIONS:
Drug: Hydrocodone Bitartrate extended-release tablet — Hydrocodone bitartrate extended-release oral tablet will be administered at a dose of 45 mg and dosed one time on Day 1. Subjects will also be dosed with naltrexone hydrochloride to block opioid effects.
  Other Names: CEP-33237

SUMMARY:
The purpose of this study is to assess the effect of varying degrees of renal impairment (mild, moderate, severe and end stage renal disease) compared with subjects with normal renal function on the pharmacokinetics of the hydrocodone bitartrate extended-release tablet.

DETAILED DESCRIPTION:
This is a multicenter, open-label, parallel-group pharmacokinetic and safety study to assess the effect of varying degrees of renal impairment (mild, moderate, severe and end stage renal disease [ESRD])on the pharmacokinetics of the hydrocodone bitartrate extended-release tablet at a single dose of 45 mg as compared with subjects with normal renal function. The study consists of a screening visit within 28 days before study drug administration (visit 1), followed by a single-dose administration period including a 144-hour pharmacokinetic sampling period (visit 2) with a final assessment after the final pharmacokinetic sample is collected or upon early withdrawal, and a follow-up visit 48 to 72 hours after the last discharge from the study center (visit 3). Subjects will be categorized into either the control group with normal renal function or one of the four groups of subjects with varying degrees of renal impairment. Up to 12 subjects in each of the 4 renal impairment groups and up to 16 subjects with normal renal function will be enrolled to achieve the targeted minimum of 8 subjects in each renal impairment group and 10 subjects with normal renal function completing the study. Eligible subjects will check in to the study center on day -1. Subjects who continue to meet the criteria for enrollment will receive a single dose of the hydrocodone bitartrate extended-release tablet on day 1. Subjects will receive one 50-mg tablet of naltrexone hydrochloride to block opioid receptors and minimize opioid related adverse events approximately 15 and 3 hours before and approximately 9 and 21 hours after study drug administration. Blood and urine samples will be collected just before study drug administration and over a 144-hour period after study drug administration. Safety will be assessed throughout the study by monitoring the occurrence of adverse events, clinical laboratory test results, vital signs measurements,12-lead ECG findings, physical examination findings, SpO2 findings, and use of concomitant medications. Subjects who complete all scheduled visits will have final procedures and assessments performed prior to discharge from the study center after pharmacokinetic sampling is complete. All subjects will be asked to return for a follow-up visit.

ELIGIBILITY:
Key Inclusion Criteria:

All subjects:

* Written informed consent is obtained.
* The subject is a man or woman at least 18 years of age, with a body mass index (BMI) of 20 kg/m2 or more.
* Women must be surgically sterile, 2 years postmenopausal, or, if of child-bearing potential, be using a medically accepted method of contraception, and agree to continued use of this method for the duration of the study and for 30 days after discontinuation of study drug.
* The subject is a nonsmoker or smokes less than 10 cigarettes per day.
* The subject's vitamin usage is stable for at least 2 weeks before study drug administration and the subject's prescription and over-the-counter (OTC) medication dosage is stable.
* The subject must be willing and able to comply with study restrictions and to remain at the clinic for the required duration of the administration period during the study.

Subjects with normal renal function:

* The subject is in generally good health as determined by medical and psychiatric history, physical examination, ECG, serum chemistry, hematology, urinalysis, and serology.
* The subject has an estimated creatinine clearance >80 mL/min.

Subjects with renal impairment:

* Subjects may have concurrent stable medical conditions in addition to renal impairment but may be included only if the investigator and protocol-specified contact for medical issues consider that the condition will not introduce an additional risk factor, and will not interfere with the study objectives and procedures (e.g., subjects with diabetes that has been stable, essential hypertension).
* Subjects are renally impaired as defined by 1 of the following categories:
* subjects with ESRD must be on hemodialysis for at least 6 months prior to enrollment and be receiving standard in-center thrice weekly treatments
* subjects with severe renal impairment must have an estimated creatinine clearance of less than 30 mL/min
* subjects with moderate renal impairment must have an estimated creatinine clearance of 30-50 mL/min
* subjects with mild renal impairment must have an estimated creatinine clearance of greater than 50 and up to 80 mL/min

Key Exclusion Criteria:

All subjects:

* The subject is a poor metabolizer of cytochrome P450 (CYP) 2D6 substrates based on genotyping performed at screening.
* The subject has used an inducer (other than weak inducers) of CYP3A4/5 or CYP2D6 within 28 days prior to study drug administration. NOTES: Topical use of a medication that is known to be an inducer of CYP3A4/5 or CYP2D6 may be permitted after consultation with the medical monitor. No medication will be permitted within 2 hours before or after study drug administration.
* The subject has used an inhibitor (other than weak inhibitors) of CYP3A4/5 or CYP2D6 within 14 days or 5 half-lives (whichever is longer) prior to study drug administration. NOTES: Topical use of a medication that is known to be an inhibitor of CYP3A4/5 or CYP2D6 may be permitted after consultation with the medical monitor. No medication will be permitted within 2 hours before or after study drug administration.
* The subject is a pregnant or lactating woman. (Any women becoming pregnant during the study will be withdrawn from the study.)
* The subject has any disorder that may interfere with drug absorption, distribution, metabolism, or excretion (including gastrointestinal surgery, excluding appendectomy). Note: Cholecystectomy performed 2 years or more prior to enrollment is permitted.
* The subject has previously participated in a study with CEP-33237.
* The subject has a known sensitivity or idiosyncratic reaction to any compound present in hydrocodone or hydromorphone, its related compounds, or to any metabolites, or naltrexone, or any compound listed as being present in a study formulation.
* The subject is unlikely to comply with the study protocol, or is unsuitable for any other reasons, as judged by the investigator.

Subjects with normal renal function:

* The subject has any clinically significant, uncontrolled medical condition (treated or untreated).
* The subject has a clinically significant deviation from normal in ECG or physical examination findings, as determined by the investigator or the protocol-specified contact for medical issues.
* Subjects with normal renal function who have a hemoglobin value of less than 12 g/dL.

Subjects with renal impairment:

* The subject has a condition that, in the opinion of the investigator or protocol-specified contact for medical issues, will introduce an additional risk factor or interfere with the study objectives and procedures.
* The subject has evidence of an unstable clinically important medical condition other than impaired renal function.
* The subject has an acute exacerbation or unstable renal function, as indicated by worsening of clinical and/or laboratory signs of renal impairment, within the 4 weeks before study drug administration.
* The subject has an acute renal disease caused by infection or drug toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | Between baseline and 144 hours following drug administration
Area under the plasma drug concentration-by-time curve (AUC) from time 0 to infinity (AUC0-∞) | Between baseline and 144 hours following drug administration

SECONDARY OUTCOMES:
Assess the safety of a single 45-mg dose of the hydrocodone bitartrate extended release tablet | Safety will be assessed from the start of study drug administration through the follow-up visit 48 to 72 hours after discharge from the study center.
  by evaluating the following:
  * occurrence of adverse events throughout the study
  * clinical laboratory (serum chemistry, hematology, and urinalysis) test results at final assessment or early withdrawal
  * vital signs measurements (blood pressure, pulse, and respiratory rate) throughout the study
  * 12-lead electrocardiogram (ECG) findings at final assessment or early withdrawal
  * physical examination findings at final assessment or early withdrawal
  * oxyhemoglobin saturation (SpO2) monitoring throughout the study
  * concomitant medication usage throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Sponsor's Medical Expert, Study Director — Cephalon, Inc.
Locations (4):
- United States (4):
  - Clinical Pharmacology of Miami, Miami, Florida
  - Orlando Clinical Research, Orlando, Florida
  - DaVita, Minneapolis, Minnesota
  - New Orleans Center, Knoxville, Tennessee